CLINICAL TRIAL: NCT07236905
Title: Improving HIV Testing Among Children Under Five in Rural Uganda
Brief Title: Improving Access to HIV Testing for Children in Uganda
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Mbarara University of Science and Technology (Other); Cornell University/Weill Cornell Medical Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R21MH135815-01 (NIH); R21MH135815-01 (NIH)
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: pediatric; child; HIV; traditional healer; Uganda; sub-Saharan Africa
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Referral and Consultation; HIV Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Healer-facilitated Test
  Interventions: Diagnostic Test: HIV saliva swab screening test
- Referral for testing (Active Comparator): Traditional healers will refer children to a nearby health center for HIV testing, which is the current standard of care.
  Interventions: Other: Referral for HIV testing

INTERVENTIONS:
Diagnostic Test: HIV saliva swab screening test — A screening swab test that can be self-administered and is commercially availble for HIV
  Arms: Intervention
Other: Referral for HIV testing — Referral by a traditonal healer to a health center for HIV testing
  Arms: Referral for testing

SUMMARY:
The goal of this study is to learn if HIV screening testing can be done for children ages 18 months to 5 years by traditional healers in Southwestern Uganda. The main questions the investigators aim to answer are:

* Will caretakers of children coming to a traditional healer for their care accept an HIV test from them?
* What views of HIV such as stigma and knowledge might affect the caretaker's choice to accept HIV testing or not for their child? Researchers will compare how many caretakers accept HIV testing for their child by a traditional healer compared to how many accept and go for testing at a nearby health center after being referred by a healer.

Participants will:

* Complete a form with the child's health history and past medical history
* Complete surveys on knowledge and understanding of HIV and stigma
* Decide to to have a rapid, oral swab test the child-participant for HIV
* Complete a follow up call once per month for 3 months to see if the child-participant went for follow up care for those in the referral group or for those who tested positive by the traditional healer

DETAILED DESCRIPTION:
Five traditional healers (TH) will be trained in the intervention to facilitate HIV counseling and testing for children under five. The other five will provide "enhanced standard of care", where healers will participate in a pre-trial educational session describing community HIV resources available for clients, and how to access them. The investigators will enroll 400 children at these 10 TH practices over a nine-month period, 200 in the intervention arm and 200 in the control. Exit interviews with all participating TH and a sample of participant caretakers will assess concepts pertinent to intervention sustainment.

RAs will arrive at the TH location within one hour to complete enrollment and written informed consent for those who endorse interest in the study after it is introduced by the TH. Once informed consent has been completed, the TH will offer counseling and rapid HIV testing or referral to the nearest health facility depending on the arm. The investigators will recruit all eligible children regardless of whether their caretaker consents for them to receive an HIV test. After enrollment, participants will receive a de-identified study identification number and caregivers will complete a locator information form with contact information (mobile phone, residency, and employment information) and information for additional contact persons. Contact persons will be peers or family members the study team can contact in case the primary caretaker is not reachable for follow-up through other means. This strategy has been feasible and effective to conduct follow up in research among adults living with HIV.

Study Training: Five participating TH for the control arm will receive a two-day training session on pediatric HIV, risk factors, and how to refer patients for testing. Five participating TH will attend a two-day training session in facilitating pediatric-specific HIV counseling and rapid oral swab testing. Both trainings will be conducted by clinicians from the ISS clinic (physicians, nurses, counselors, and social workers). Training will follow the approach in our previously effective trial, tailored to the pediatric population. A final training curriculum will be developed in Aim 1. TH will receive instruction on delivering family-centered pre-and post-HIV test counseling with observed practice sessions and hands-on use of Oraquick® oral swab test kits. These tests are endorsed by the Ugandan MoH and WHO for community layperson HIV self-testing in non-clinical settings. The test is rated as 99.3% sensitive and 99.8% specific. Verbal assessments of knowledge with teach back will occur one-on-one in a private setting. Incorrect answers will be re-explained, then assessments re-administered. Counselling and testing will be directly observed by Dr. Nansera and ISS clinicians to ensure HCT is delivered as instructed.

Study Procedures: A trained, study RA will collect demographics from the child's caretaker on enrollment including age, sex, birth history, prior HIV testing, household characteristics (income, distance to TH, mode of transportation), and biological parent data including age, marital status, and HIV history (including prior testing). RAs will administer validated scales at enrollment to measure caretaker characteristics including social support, self-efficacy, HIV-related stigma, and HIV knowledge. All scales have been validated in similar East African populations. Following informed consent by caregivers, TH will offer pre-test counseling and - if accepted - facilitate HIV testing or refer to a nearby facility depending on the arm. Method of oral swab collection will depend on caretaker and child preference: TH can perform the oral mucosal swab, or supervise caretakers in performing the swab. Counseling and testing will take place in a private location. Results are available in 15 minutes and will be delivered verbally to the caretaker and in written format. Infants less than 18 months old are not eligible to receive rapid HIV testing per MoH guidelines. Caretakers of infants will be given a referral form and instructed to go to a local clinic for HIV testing if the child has not received an HIV test in the past three months And is potentially exposed, similar to those in the control arm.

Caretakers of children with reactive tests at the TH will receive pediatric-specific post-test counseling on their child's potential diagnosis and a referral form with location and contact information for the ISS Maternal and Pediatric clinic and other nearby HIV clinics, with instructions to present to the nearest clinic for confirmatory testing as soon as possible. TH will also offer oral swab testing to biologic parents of HIV-reactive children. Caretakers of participants with non-reactive tests will receive counseling on HIV prevention strategies including primary HIV prevention for the mother and need for repeat HIV testing every three months while breastfeeding. Those at the control sites will undergo testing at the local health facility and post-test counseling per the Ugandan MOH protocol. Study staff will conduct drop-ins throughout the study and contact TH weekly to observe and answer questions about counseling, test kit use, or eligibility screening to ensure integrity and minimize social harm. Testing kits will be provided by the study for all participating TH and provided to clients at no charge. Intervention delivery will be monitored by the Project Manager using the fidelity and feedback plan developed in Aim 1.

All participants will be contacted by phone once per month for a period of three months to inquire about subsequent testing, confirmation of initial result if HIV reactive, and linkage to care and initiation of treatment for those who are confirmed as HIV positive. Caretaker-reported data will be confirmed through verification of treatment dates listed on HIV treatment cards provided those in HIV care. The investigators will also ask the participant to name their clinic; with their consent, an RA will go to that clinic to validate linkage to care and ART initiation, an approach the investigators have used in prior work. If needed, participants may be followed up in-person at their home if participants are unable to be reached by phone.

Exit Interviews will be conducted with the 5 TH in the intervention arm, and a sample of 20 participant caretakers of children enrolled at these sites, following the procedures described in Aim 1. Again, the investigators will use purposive sampling to select caretakers who represent the range of participant age, gender, HIV test results, and secondary outcomes. Interview guides will include questions that consider implementation inner (adequacy of intervention support and resources) and outer contexts (fit with national HIV priorities, potential funding sources), bridging (collaborations between TH and clinics) and innovation factors (accessibility, acceptability, and potential barriers to sustainability), and will assess any emotional distress endured during the process. Spot interviews will occur immediately after testing in an initial sample of 10 caretakers of both HIV reactive and non-reactive children within the first two weeks of the study at to assess post-test counseling adequacy, safety concerns, and any potential for social harm. All of these interviews will be audio recorded, translated, and transcribed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 months to 5 years old
* Have a parent or caregiver present who can provide informed consent
* Not previously tested for HIV in the past three months
* Npt previously known to be HIV-infected.

Exclusion Criteria:

* unwilling or unable to participate in study procedures or provide written informed consent.

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete HIV testing | from enrollment up to 3 months post
  Total number of participants who complete HIV testing

SECONDARY OUTCOMES:
Number of children with a positive HIV test | enrollment to 3 months post
  number of children who test positive for HIV
Number of HIV-positive children who initiate antiretroviral treatment (ART) | enrollment to 3 months post
  number of HIV positive children who initiate ART

CONTACTS AND LOCATIONS:
Overall Officials: Anneka Hooft, MD, MPH, Principal Investigator — University of California, San Francisco; Radhika Sundararajan, MD, PhD, Principal Investigator — Weill Cornell School of Medicine; Denis Nansera, MD, Principal Investigator — Mbarara University of Science and Technology
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be deposited in the NIMH Data Archive as required by the funders. Data dictionaries and descriptions will be provided. Data will be deidentified prior to deposition.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months after publication of results with no end date (or as determined by NDA)
Access Criteria: Access will be moderated by NDA with those fulfilling requirements having access to data
URL: https://nda.nih.gov/nda/access-data-info

REFERENCES:
- Available data/document: Individual Participant Data Set — https://nda.nih.gov/nda/access-data-info — data is not yet available but will be added to respository once acquired.